CLINICAL TRIAL: NCT07001150
Title: Clinical Study Evaluating the Possible Role of Silymarin in Neuroprotection and Symptom Management in Parkinson's Disease
Brief Title: Role of Silymarin in Neuroprotection and Symptom Management in Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Prof. Sahar Kamal Hegazy,Head of Clinical Pharmacy Department,Faculty of Pharmacy,Tanta University (Unknown); Dr. Raed Ahmed Abdel-Maboud,Lecturer of neurology,Faculty of Medicine,Tanta University (Unknown)
Responsible Party: Principal Investigator, Nour Amr Ahmed Mosaad Elsherbeny, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1331999
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Silymarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): 25 patients who will receive their standard dopamine replacement therapy for 6 months
  Interventions: Drug: levodopa-carbidopa
- Silymarin group (Active Comparator): 25 patients who will receive their standard dopamine replacement therapy plus silymarin 140mg three times daily for 6 months
  Interventions: Drug: levodopa-carbidopa; Drug: Silymarin

INTERVENTIONS:
Drug: levodopa-carbidopa — Carbidopa/levodopa is a combination of two medications: carbidopa and levodopa. It is primarily used to manage the symptoms of Parkinson's disease. The main and most effective treatment strategy for motor symptoms in Parkinson's disease relies on replenishing dopamine levels through the use of L-dopa.
Drug: Silymarin — Silymarin, a polyphenolic flavonoid renowned for its potent antioxidant properties, is employed clinically for managing hepatic disorders. Its antioxidant effects are primarily attributed to its ability to scavenge free radicals.
  Arms: Silymarin group

SUMMARY:
Parkinson's disease (PD) is a leading neurodegenerative movement disorder, marked by a gradual loss of dopamine-producing neurons in the substantia nigra pars compacta (SNpc) and the accumulation of α-synuclein protein aggregates. Silymarin, a polyphenolic flavonoid renowned for its potent antioxidant properties, will be studied for its neuroprotective effects in PD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 65 years old
* Both sexes
* Patients with Parkinson's disease on dopamine replacement therapy
* Modified Hoehn and Yahr stage, MHY 1-4 (29)

Exclusion Criteria:

* Subjects < 18 years of age
* Pregnant or breastfeeding women
* Suspected hypersensitivity to silymarin or multivitamins
* Advanced liver disease (e.g., ascites, bleeding esophageal varices, and hepatic encephalopathy)
* Subjects with morbid obesity, i.e., a Body Mass Index (BMI) > 40
* Subjects with severe illness, e.g., multisystem failure, cancer, or poorly controlled diabetes, i.e., known diabetic with Hemoglobin A1C (HbA1C)>7%
* Current use of Silymarin or recent use within the past two weeks.
* Other conditions, which, in the opinion of the investigators, make the patient unsuitable for enrollment.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | 6 months
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a rating tool used to determine the severity and progression of Parkinson's disease in patients

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Hospital for Mental Health, Tanta, Tanta, Qism 2, Egypt

IPD SHARING:
Plan to Share IPD: No